CLINICAL TRIAL: NCT02151500
Title: Stress and Health Interview for Primary Care Patients With Medically Unexplained Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark A. Lumley, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSU.HIC.036514B3E
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Somatoform Disorders
Keywords: Medically Unexplained Symptoms (MUPS); Somatoform disorders; Chronic pain; Somatic symptoms; Emotional processing; Primary Care
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress and Health Interview (Experimental): Stress and Health Interview is an experiential assessment technique
  Interventions: Behavioral: Stress and Health Interview
- Wait-list Control (No Intervention): Standard medical care until the 6-week follow-up is completed

INTERVENTIONS:
Behavioral: Stress and Health Interview — A stress and health interview which aims to help patients: a) disclose their stressful experiences and emotional conflicts, which might be contributing to their symptoms; b) learn about associations between their stress and physical symptoms; and c) learn about the potential value of experiencing and expressing their emotions related to these stressful situations.
  Arms: Stress and Health Interview

SUMMARY:
The goal of this study is to test the feasibility and acceptability of providing an experiential assessment interview that targets emotional and stressful experiences in primary care. In this randomized, controlled trial, the investigators will compare an interview condition to a wait-list control condition. The investigators hypothesize that helping individuals first identify the links between their stress and symptoms will likely increase their awareness and endorsement of the link between stress and physical symptoms, including a willingness to engage in stress management techniques. It is also expected that helping raise an individual's awareness about their symptoms, followed by an experience and expression of unexpressed emotions is likely to influence their physical symptoms and psychological status.

DETAILED DESCRIPTION:
Emotional stress, particularly when a patients inhibits their experiences and feelings, contributes to physical symptoms. However, primary care patients with medically unexplained symptoms are rarely assessed for the stress and emotions in an comprehensive manner. The goal of this study is to test the feasibility and acceptability of providing an experiential assessment interview that targets emotional and stressful experiences in primary care with medically unexplained physical symptoms. In this randomized, controlled trial, the investigators will compare an interview condition to a wait-list control condition. The interview will review patients health history, psychosocial history, make links between the two, and help patients identify and express emotions related to conflicts or victimization. The investigators hypothesize that helping individuals first identify the links between their stress and symptoms will likely increase their awareness and endorsement of the link between stress and physical symptoms, including a willingness to engage in stress management techniques. It is also expected that helping raise an individual's awareness about their symptoms, followed by an experience and expression of unexpressed emotions is likely to influence their physical symptoms and psychological status.

ELIGIBILITY:
Inclusion Criteria:

* Participants must score above 10 (moderate range) on the Patient Health Questionnaire-15, which is a measure of a range of medical symptoms that are often medically unexplained.

Exclusion Criteria:

1. Conditions that could interfere with the interview:

   * non-English speaking
   * psychosis
   * dementia
   * mental impairment
2. The presence of disease or injury that could account for the physical symptoms. - Examples: autoimmune disease, bodily injury, serious infection, cancer, heart disease, COPD, post-stroke.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Symptom Interpretation Questionnaire (SIQ) | Change from baseline symptom attribution at 6-weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire-15 (PHQ-15) | Change from baseline in symptom severity at 6-weeks
Brief Pain Inventory (BPI) | Change from baseline pain at 6-weeks
Brief Symptom Inventory (BSI) | Change from baseline symptoms at 6-weeks
Insomnia Severity Scale (ISI) | Change from baseline insomnia at 6-weeks
Brief Fatigue Inventory | Change from baseline fatigue at 6-weeks
Satisfaction with Life Scale (SWLS) | Change from baseline life satisfaction at 6-weeks
Emotional Approach Coping Scale (EAC) | Change from baseline emotional approach coping at 6-weeks
Emotional Processing Scale (EPS) | Change from baseline emotional processing at 6-weeks
Inventory of Interpersonal Problems Scale (IIP-32) | Change from baseline interpersonal problems at 6-weeks
Pain Catastrophizing Scale (PCS) | Change from baseline pain catastrophizing at 6-weeks
Change Assessment Questionnaire | Changes from baseline stage of change at 6-weeks
McGill Pain Questionnaire (SF-MPQ-2) | Change from baseline pain at 6-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Lumley, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University Family Medicine Clinic, Rochester Hills, Michigan, United States

REFERENCES:
- [Derived] Ziadni MS, Carty JN, Doherty HK, Porcerelli JH, Rapport LJ, Schubiner H, Lumley MA. A life-stress, emotional awareness, and expression interview for primary care patients with medically unexplained symptoms: A randomized controlled trial. Health Psychol. 2018 Mar;37(3):282-290. doi: 10.1037/hea0000566. Epub 2017 Nov 20. PMID 29154608